CLINICAL TRIAL: NCT01038986
Title: A Post-marketing Multi-center Observational Study to Provide Data Describing the Safety and Effectiveness of CUREXCELL™ as it is Applied in a Real-life Setting for Treatment in Patients With Chronic and/or Refractory Wounds
Brief Title: A Post-marketing Observational Study of Cell Therapy for Chronic Wounds
Status: Completed | Type: Observational
Sponsor: Macrocure Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MC101-IL-01
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Wounds
Keywords: chronic wound; refractory wound; CureXcell; activated cell suspension
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CureXcell treated: Patients with chronic and/or refractory wounds for at least 4 weeks with no improvement that have been referred by their physician for CureXcell treatment
  Interventions: Biological: CureXcell

INTERVENTIONS:
Biological: CureXcell — The CureXcell™ dosage form consists of an aseptically-processed activated cell suspension that has been isolated, activated and purified from the peripheral blood of healthy allogeneic donors, by hypo-osmotic shock, using the MacroCure custom closed bag system.

SUMMARY:
A post-marketing multi-center observational study to provide data describing the safety and effectiveness of CUREXCELL™ as it is applied in a real-life setting for treatment in patients with chronic and/or refractory wounds.

DETAILED DESCRIPTION:
Chronic wounds can be categorized into two main groups: (a) chronic ulcers, such as diabetic foot ulcers, venous leg ulcers and pressure (decubitus) ulcers (b) post-operative or traumatic, difficult-to-heal wounds, some of which may be infected such as sternal wound infections following cardiac surgery or wounds following abdominal or orthopedic surgery. Age, peripheral vascular disease, infection, diabetes mellitus, auto-immune dis., obesity, cardiac disease, cardiac failure, malnutrition, immunological deficiencies, steroid treatment, bed confinement and prolonged operation time are among the causes of wound repair delay or failure and often results in considerable morbidity and mortality. In addition, these wounds lengthen hospital stays, significantly increase the cost of care, and negatively impact the quality of life of both the patients and care giversCurrently available wound care products include various dressings, ointments, gels, antiseptic agents and devices. These products are intended to supply a suitable environment for wound healing (e.g. moist environment, particular factors required for the healing process), but they do not provide an adequate solution for this growing problem of chronic wounds.

Macrocure has developed an advanced cellular therapy for wound healing named Curexcell™. Curexcell™ not only provides the natural environment for wound healing, but also ensures that the appropriate cell activities and factor secretions are maintained as required during each of the stages of wound healing. The product contains primed/activated Monocytes, Neutrophils and Lymphocytes derived from whole blood unit, which are key role players in the normal natural wound healing process. The cells are injected locally into the wound bed.

The proposed study is a post-marketing observational study (PMOS) in which the decision to use Curexcell™ for treatment of patients with chronic and/or refractory wounds are made by local physicians. Curexcell™ will be administered to the patient in accordance with the Instructions for Use.

In this PMOS, there is no control by the investigator with respect to patients, duration and frequency of follow-up and the method by which patients are managed in general. This design truly reflects real-life circumstances.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic and/or refractory wounds that have been referred by their physician for CUREXCELLTM treatment
* Signed consent form

INCLUSION CRITERIA FOR THE BLINDING GUESSING TEST

* Patients with chronic lower extremity ulcers (on malleoli and below) and diabetes mellitus
* Signed the blinding guessing test section of the consent form
* Were not treated in the past by CureXcell

Exclusion Criteria:

* Patients with known or suspected present malignancy (except for successfully treated basal cell carcinoma) within the past 3 years.
* Patients with gangrene
* Patients for whom amputation or a complete resection of the infection site is planned component of treatment
* Patients simultaneously participating in any interventional clinical trial
* Patients with any other known or suspected condition that may jeopardize adherence to registry protocol requirements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic and/or refractory wounds that have been referred by their physician for CureXcell treatment
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2009-12; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Incidence and frequency of adverse experiences | 3 years

SECONDARY OUTCOMES:
Percent of complete healing following CureXcell™ treatments | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Itzchak Zivner, MD, Principal Investigator — Sheba Medical Center; Eli Peled, M.D., Principal Investigator — Rambam Health Care Campus, Israel; Dean David Ad-El, M.D., Principal Investigator — Rabin-Schnider Medical Center
Locations (3):
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Tel Litwinsky

REFERENCES:
- [Background] Leor J, Rozen L, Zuloff-Shani A, Feinberg MS, Amsalem Y, Barbash IM, Kachel E, Holbova R, Mardor Y, Daniels D, Ocherashvilli A, Orenstein A, Danon D. Ex vivo activated human macrophages improve healing, remodeling, and function of the infarcted heart. Circulation. 2006 Jul 4;114(1 Suppl):I94-100. doi: 10.1161/CIRCULATIONAHA.105.000331. PMID 16820652
- [Background] Orenstein A, Kachel E, Zuloff-Shani A, Paz Y, Sarig O, Haik J, Smolinsky AK, Mohr R, Shinar E, Danon D. Treatment of deep sternal wound infections post-open heart surgery by application of activated macrophage suspension. Wound Repair Regen. 2005 May-Jun;13(3):237-42. doi: 10.1111/j.1067-1927.2005.130304.x. PMID 15953041
- [Background] Zuloff-Shani A, Kachel E, Frenkel O, Orenstein A, Shinar E, Danon D. Macrophage suspensions prepared from a blood unit for treatment of refractory human ulcers. Transfus Apher Sci. 2004 Apr;30(2):163-7. doi: 10.1016/j.transci.2003.11.007. PMID 15062757
- [Background] Frenkel O, Shani E, Ben-Bassat I, Brok-Simoni F, Rozenfeld-Granot G, Kajakaro G, Rechavi G, Amariglio N, Shinar E, Danon D. Activated macrophages for treating skin ulceration: gene expression in human monocytes after hypo-osmotic shock. Clin Exp Immunol. 2002 Apr;128(1):59-66. doi: 10.1046/j.1365-2249.2002.01630.x. PMID 11982591
- [Background] Danon D, Kowatch MA, Roth GS. Promotion of wound repair in old mice by local injection of macrophages. Proc Natl Acad Sci U S A. 1989 Mar;86(6):2018-20. doi: 10.1073/pnas.86.6.2018. PMID 2928316